CLINICAL TRIAL: NCT03600051
Title: Phonokardiographie Bei Erwachsenen
Brief Title: Automated Phonocardiography Analysis in Adults
Status: Completed | Type: Observational
Sponsor: CSD Labs GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: GRZ03 (PbE)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Aortic Insufficiency; Aortic Stenosis; Mitral Insufficiency; Mitral Insufficiency and Aortic Stenosis; Tricuspid Regurgitation; Insufficiency, Pulmonary; Insufficiency, Tricuspid
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Automated Heart Murmur Detection AI — Automated AI algorithm-based analysis of digital heart sound recordings to detect pathological heart murmurs. Heart sound recordings were fully blinded before undergoing one-time automated analysis. Algorithm results for each recording included: AHA classification (I "pathologic" versus III "innocent/no murmur"), murmur timing, murmur grade, heart rate and S1/S2 identification.

SUMMARY:
Background: Computer aided auscultation in the differentiation of pathologic (AHA class I) from no- or innocent murmurs (AHA class III) via artificial intelligence algorithms could be a useful tool to assist healthcare providers in identifying pathological heart murmurs and may avoid unnecessary referrals to medical specialists.

Objective: Assess the quality of the artificial intelligence (AI) algorithm that autonomously detects and classifies heart murmurs as either pathologic (AHA class I) or as no- or innocent (AHA class III).

Hypothesis: The algorithm used in this study is able to analyze and identify pathologic heart murmurs (AHA class I) in an adult population with valve defects with a similar sensitivity compared to medical specialist.

Methods: Each patient is auscultated and diagnosed independently by a medical specialist by means of standard auscultation. Auscultation findings are verified via gold-standard echocardiogram diagnosis. For each patient, a phonocardiogram (PCG) - a digital recording of the heart sounds - is acquired. The recordings are later analyzed using the AI algorithm. The algorithm results are compared to the findings of the medical professionals as well as to the echocardiogram findings.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a heart defect verified by echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly in-patient subjects admitted to the Division of Cardiology, University Hospital Graz, Austria. All patients had known pathological murmurs caused by multiple valve defects, confirmed by gold standard echocardiography. Defects were interpreted by the cardiologist as "low, medium or high" severity. Altogether, 155 valve defects were observed, including insufficiencies of the aortic, mitral, tricuspid, and pulmonary valves; and stenosis of the aortic and mitral valves.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity for pathological heart murmur detection | 2 months
  Ability to detect a pathological heart murmur in digital heart sound recordings obtained from an elderly population with heart valve disease.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Riedlbauer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- University Hospital, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No